CLINICAL TRIAL: NCT07261098
Title: A Prospective Study of the Efficacy and Safety of Angiotensin Receptor-neprilysin Inhibitor in Patients With Advanced Lung Cancer and Concurrent Hypertension
Brief Title: The Efficacy and Safety of ARNI on the Outcome of Advanced Lung Cancer With Concurrent Hypertension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Liang Zhao, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025IIT-ARNI-0001
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lung Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The patients of this cohort take anti-hypertensive medicine other than ARNI, such as angiotensin receptor blockers, calcium channel blockers, and diuretics.
  Interventions: Drug: Anti-hypertensive drugs except ARNI
- ARNI group (Experimental): The patients of this cohort take ARNI as anti-hypertensive medicine.
  Interventions: Drug: ARNI

INTERVENTIONS:
Drug: ARNI — ARNI is prescribed for lung cancer patients with concurrent arterial hypertension
  Arms: ARNI group
Drug: Anti-hypertensive drugs except ARNI — Anti-hypertensive drugs except ARNI
  Arms: Control group

SUMMARY:
Despite the rapid development of novel anti-cancer therapeutic agents and ensuing improved prognosis, lung cancer remains the leading cause of cancer-related death globally, of which the majority of mortality could be attributed to advanced lung cancer. Hypertension is frequently diagnosed among patients with advanced lung cancer, either a comorbidity or complication, and is associated with increased incidence of cardiac adverse events, such as heart failure, coronary artery disease, and cardiac arrhythmias, hence aggravating patients' prognosis.

Sacubitril/valsartan, a combination of an angiotensin II receptor blocker and neprilysin inhibitor (ARNI), is a novel agent to treat HF and has been approved to treat hypertension in China, of which the cardio-protective effect has been widely acknowledged. Yet current knowledge remains lacking on the influence of ARNI on the prognosis of advanced lung cancer with concurrent hypertension. The present study aimed to investigate the prognostic value of ARNI in patients with advanced lung cancer and concurrent hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent (ICF) and able to understand and comply with the study requirements and assessment schedule.
* Male or female aged ≥18 years and < 80years at the time of signing the ICF.
* Histologically or cytologically confirmed advanced lung cancer (TNM III-TNM IV) based on the 8th edition of the AJCC staging system
* Patients were diagnosed hypertension before the diagnosis of advanced lung cancer
* ECOG performance status score ≤ 1.
* Adequate organ function during the screening period

Exclusion Criteria:

* Predicted survival period less than 12 months
* Female patients if pregnant.
* Hypersensitivity to any component of ARNI
* Severe renal dysfunction (eGFR<30ml/min/1.73m2)
* Severe liver dysfunction (Child-Pugh C)
* Bilateral renal artery stenosis or solitary renal artery stenosis
* Refractory hyperkalemia
* Moderate or severe aortic stenolsis
* Obstructive hypertrophic cardiomyopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | From enrollment to the end of treatment at 24 months
  Patients deceased during follow-up regardless of the cause.

SECONDARY OUTCOMES:
Major adverse cardiovascular event | From enrollment to the end of treatment at 24 months
  Major adverse cardiovascular events include cardiovascular death, hospitalization due to heart failure, acute coronary syndrome, and myocardial infarction.